CLINICAL TRIAL: NCT06719089
Title: Evaluation of the Safety and Performance of the Hydrustent® Biodegradable Hydrogel Ureteral Stent in Patients With Nephrolithiasis: A Multicentric, Randomized, Controlled Study
Brief Title: Evaluation of the Safety and Performance of the Hydrustent® Biodegradable Hydrogel Ureteral Stent
Acronym: Hydrustent
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hydrumedical (Industry)
Collaborators: Blueclinical, Ltd. (Other); Clinical Academic Center (2CA-Braga) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hydrustent
Record Dates: First submitted 2024-10-04; First posted 2024-12-05 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Urinary Lithiasis
Keywords: Biodegradable ureteral stent; kidney stones; Hydrustent; Hydrumedical
MeSH Terms: conditions — Urolithiasis; Kidney Calculi

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Investigators that will place the stent will not be the same that will perform the follow-up visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rocamed RocaJJ Soft (Active Comparator)
  Interventions: Device: PolyUrethane Double Loop Ureteral Stent
- Hydrustent® (Experimental)
  Interventions: Device: Biodegradable double loop ureteral stent

INTERVENTIONS:
Device: Biodegradable double loop ureteral stent — This ureteral stent is based on natural polymers and degrades inside the human body without causing obstruction, avoiding the need of a second surgery for stent removal and minimizing complications related to encrustation and bacterial infections.
  Arms: Hydrustent®
Device: PolyUrethane Double Loop Ureteral Stent — This ureteral stent is a double J made of 100% polyurethan, heat-sensitive and radiopaque for excellent patient tolerance and high incrustation resistance.
  Arms: Rocamed RocaJJ Soft

SUMMARY:
The goal of this clinical investigation is to evaluate whether the Hydrustent® medical device is safe and if maintain the urinary flow inside the ureter in adults.

The main questions it aim to answer are:

* Does Hydrustent® maintain urinary patency post-surgery in adults?
* What medical issues do participants experience while using Hydrustent®?

Researchers will compare the Hydrustent® medical device to a comparator (a standard medical device used in clinical practice) to determine whether Hydrustent® is at least non-inferior in terms of safety and efficacy.

Other questions that the study will answer are:

* Does Hydrustent® exhibit a durability of at least 24 hours?
* Does Hydrustent® prevents the need of the surgical procedure to remove the ureteral stent?
* Does Hydrustent® reduce urinary symptoms associated with a ureteral stent?

Participants will:

* Have either the Hydrustent® or a comparator device inserted following the removal of ureteral or renal stones via endourological techniques.
* Be monitored for 3 months post-surgery through regular follow-up visits.
* Complete questionnaires and undergo imaging exams, as well as blood and urine analyses to assess recovery.

DETAILED DESCRIPTION:
Multicentric, randomized, controlled clinical study comprising both phases of the pre-market device clinical development stage: pilot and pivotal. The first exploratory phase of the study (16 participants) will assess the safety of Hydrustent® for the first time in humans, while providing preliminary results on its efficacy. Following this, the second phase is confirmatory (118 participants), allowing the collection of the information necessary to evaluate the clinical performance and safety of Hydrustent®.

ELIGIBILITY:
Pilot phase:

Inclusion:

* Subjects with the ability to understand the requirements of the study, who have provided written ICF before any assessment is performed, and are willing to undergo all FU assessments according to the specified schedule;
* Adult patients, males or females, aged between 18 and 70 years old;
* Subjects with ureteral and/or renal stones who have undergone a successful, uncomplicated, unilateral URS and RIRS, with clinical indication to place a post-operative US, as judged by the medical investigator;
* Subjects with a height and body sizeable to accommodate a 22, 24, 26, 27 and 28 cm long US and diameter of 7 Fr, as judged by the medical investigator;
* Female participants of childbearing potential and male participants whose partner is of childbearing potential must be willing to ensure that they or their partner use protocol's recommended effective contraception methods during all the trial duration;
* Male participants must agree to refrain from donation of semen from the start of the study treatment up to the end of the study.

Exclusion:

* Subjects with urinary anatomic malformations or previous relevant surgical modifications.
* Subjects with known/suspicion of urothelial or renal tumour;
* Subjects with known/suspicion of extrinsic compression of the ureter and/or stricture;
* Subjects with known/suspicion of ureteral perforation and/or fistula;
* Subjects under active treatment for bladder outlet obstruction (e.g., benign prostatic obstruction), neurogenic bladder, overactive bladder, and/or urge urinary incontinence;
* Subjects with a solitary kidney;
* Subjects with calculated GFR below 60 mL/min/1.73m2;
* Subjects with known renal insufficiency or chronic impairment;
* Subjects with post-operative suspicion/known incomplete stone fragmentation with the presence of relevant residual urinary lithiasis, requiring an additional procedure;
* Subjects with active history of bleeding diathesis or currently taking anticoagulants (except antiplatelet agents);
* Subjects with pre-operative evidence of staghorn calculi;
* Subjects with suspicious/diagnosed UTI at the time of US placement, or pre-operative positive urine culture or active UTI taking antibiotic medication;
* Subjects with contrast allergy; Pregnant, lactating, or women of childbearing potential who do not employ a highly effective contraceptive method as judged by the medical investigator, and/or who are not willing to use a highly effective contraception for the duration of study participation;
* Subject with a known severe psychiatric disorder, substance abuse, or other reason for being unable to follow study FU instructions or unable to reliably complete patient questionnaires;
* Subjects with signs of local or systemic acute/active or chronic infections;
* Subjects with sensibility or known hypersensitivity to the implantable materials;
* Subjects with ureteral blockage or stricture;
* Subjects with failed guidewire placement or failed ureteroscopy access;
* Subjects with suspect ureteral avulsion;
* Subjects with untreated infected urinary obstruction of the kidneys (pyonephrosis);
* Subjects with vascular abnormalities of the renal pelvis outlet;
* Subjects with unexplained haematuria;
* Subjects with significant urethral obstruction;
* Subjects with concomitant or untreated bladder lithiasis;
* Any other condition that would deem a subject ineligible for treatment with the investigational device in the opinion of the medical investigator;
* Subject is known to be currently enrolled in another investigational study.

Pivotal phase:

Inclusion:

* Subjects with the ability to understand the requirements of the study, who have provided written or oral informed consent form before any assessment is performed, and are willing to undergo all FU assessments according to the specified schedule;
* Adult patients, males or females, aged > 18 years old;
* Subjects with ureteral and/or renal stones who have undergone a successful, unilateral ureteroscopy and retrograde intra-renal surgery, with clinical indication to place a post-operative US, as judged by the medical investigator;
* Subjects with a height and body sizeable to accommodate a 22, 24, 26, 27 and 28 cm long US and diameter of 7 Fr, as judged by the medical investigator;
* Female participants of childbearing potential and male participants whose partner is of childbearing potential must be willing to ensure that they or their partner use protocol's recommended effective contraception methods during all the trial duration;
* Male participants must agree to refrain from donation of semen from the start of the study treatment up to the end of the study.

Exclusion:

* Urinary anatomic malformations or previous relevant surgical modifications;
* Subjects with known/suspicion of urothelial or renal tumour;
* Subjects with known/suspicion of extrinsic compression of the ureter and/or stricture;
* Subjects with known/suspicion of ureteral perforation and/or fistula;
* Subjects under active treatment for bladder outlet obstruction (e.g., benign prostatic obstruction), neurogenic bladder, overactive bladder, and/or urge urinary incontinence;
* Subjects with a solitary kidney;
* Subjects with calculated Glomerular Filtration Rate below 60 mL/min/1.73m2;
* Subjects with post-operative suspicion/known incomplete stone fragmentation with the presence of relevant residual urinary lithiasis, requiring an additional procedure;
* Subjects with active history of bleeding diathesis or currently taking anticoagulants (except antiplatelet agents);
* Subjects with pre-operative evidence of staghorn calculi;
* Subjects with suspicious/diagnosed urinary tract infection at the time of ureteral stent insertion, or pre-operative positive urine culture or active urinary tract infection taking antibiotic medication;
* Subjects with contrast allergy;
* Pregnant, lactating, or women of childbearing potential who do not employ a highly effective contraceptive method and/or who are not willing to use a highly effective contraception for the duration of study participation;
* Subject with a known severe psychiatric disorder, substance abuse, or other reason for being unable to follow study FU instructions or unable to reliably complete patient questionnaires;
* Subjects with signs of local or systemic acute/active or chronic infections;
* Subjects with sensibility or known hypersensitivity to the implantable materials;
* Subjects with ureteral blockage or stricture;
* Subjects with failed guidewire placement or failed ureteroscopy access;
* Subjects with suspect ureteral avulsion;
* Subjects with untreated infected urinary obstruction of the kidneys (pyonephrosis);
* Subjects with vascular abnormalities of the renal pelvis outlet;
* Subjects with unexplained haematuria;
* Subjects with significant urethral obstruction;
* Subjects with concomitant or untreated bladder lithiasis;
* Any other condition that would deem a subject ineligible for treatment with the investigational device in the opinion of the medical investigator;
* Subject is known to be currently enrolled in another investigational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint assessed through adverse events and device deficiencies (Pilot and pivotal phases) | From surgery to the end of treatment at day 28
  Evaluation of the number, severity, and intensity of AEs and DDs at least possibly related to either the investigational device or the comparator device that occurred within 28±1 days of stent placement.
Primary efficacy outcome assessed by the urine drainage after stent placement (Pivotal phase) | From surgery to day 1
  Urine patency will be assessed using a composite endpoint based on the following criteria:
  1. Diuresis (range within 0.5 to 1.5 mL/kg/h).
  2. Creatinine levels in blood tests (range within 0.7 to 1.2 mg/dL for men and 0.5 to 1.0 mg/dL for women).
  3. CT scan to assess the adequate upper urinary tract urine drainage (defined as the absence of significative hydronephrosis)
  4. Lack of surgical intervention in the stented ureter.

SECONDARY OUTCOMES:
Overall clinical success (efficacy) by evaluating the urine drainage after stent placement (Pilot phase) | From surgery to the end of treatment at day 28
  Urine patency will be assessed using a composite endpoint based on the following criteria:
  1. Diuresis (range within 0.5 to 1.5 mL/kg/h).
  2. Creatinine levels in blood tests (range within 0.7 to 1.2 mg/dL for men and 0.5 to 1.0 mg/dL for women).
  3. CT scan to assess the adequate upper urinary tract urine drainage (defined as the absence of significative hydronephrosis)
  4. Lack of surgical intervention in the stented ureter.
Overall clinical success by evaluating the urine drainage after stent placement (Pivotal phase) | From surgery to the end of treatment at day 28
  Urine patency will be assessed using a composite endpoint based on the following criteria:
  1. Creatinine levels in blood tests (range within 0.7 to 1.2 mg/dL for men and 0.5 to 1.0 mg/dL for women).
  2. CT scan to assess the adequate upper urinary tract urine drainage (defined as the absence of significative hydronephrosis)
  3. Lack of surgical intervention in the stented ureter.
Overall safety assessed through adverse events and device deficiencies (Pilot and pivotal phases) | From surgery to the end of study at day 90
  Evaluation of the number, severity, and intensity of AEs at least possibly related to the devices occurring and number, type and severity of DDs.
Assessment of the durability of the experimental device (Pilot and pivotal phases) | Day 1
  Presence of an intact device with no radiographic evidence of breakage or dissolution assessed by radiological assessment
Technical success of the experimental device (Pilot and pivotal phases) | Day 28
  Complete degradation of the investigational stent as measured by radiological assessment (CT scan).
Devices tolerability through the assessment of urinary symptoms (Pilot and pivotal phases) | Screening phase, during the treatment phase and up to the end of the study at day 90
  Assessment of urinary symptoms via the Ureteral Stent Symptom Questionnaire (USSQ).
  The total score of the questionnaire is the sum of all items across the following symptom sections: urinary symptoms, pain, sexual issues, general health, and work performance. A higher total score reflects a greater burden of symptoms and worse quality of life.
Devices tolerability through the assessment of urinary symptoms (Pilot and pivotal phases) | Screening phase, during the treatment phase and up to the end of the study at day 90
  Assessment of urinary symptoms via the Visual Analog Scale (VAS). Study participants mark their symptom intensity on a continuous line 10 centimetres long, the extremes of which indicate "no pain" and "maximum pain". A higher score indicates greater pain intensity.
Devices tolerability through the assessment of urinary symptoms (Pilot and pivotal phases) | During the treatment phase and up to the end of the study at day 90
  Assessment of urinary symptoms via the need of pain medication. If intervention for pain management is required, it suggests that the urinary symptoms are more severe.
Devices tolerability through the assessment of urinary symptoms (Pilot and pivotal phases) | Screening phase, during the treatment phase and up to the end of the study at day 90
  Assessment of urinary symptoms via the International Index of Erectile Function (IIEF-5) for male participants.
  The 5-item tool, with each item scored from 1 to 5, generates a total score ranging from 5 to 25 points. Lower scores indicate poorer sexual functioning, while higher scores reflect better erectile functioning.
Devices tolerability through the assessment of urinary symptoms (Pilot and pivotal phases) | Screening phase, during the treatment phase and up to the end of the study at day 90
  Assessment of urinary symptoms via the International Prostate Symptom Score (IPSS) for male participants.
  The questionnaire consists of two sections: fhe first section includes a 7-item tool, with each item scored from 0 to 5, generating a total score ranging from 0 to 35 points. The second section assesses quality of life, with scores ranging from 0 to 6. Lower scores indicate fewer urinary symptoms and better quality of life related to urinary symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Coordinating Investigator, Study Chair — Paulo Mota
Locations (4):
- Portugal (4):
  - Unidade Local de Saúde da Região de Aveiro (ULSRA), E.P.E., Aveiro, Aveiro District
  - Unidade Local de Unidade Local de Saúde do Alto Ave (ULSAAVE), E.P.E, Guimarães, Braga District
  - Hospital CUF Tejo, Lisbon
  - Unidade Local de Saúde do Alto Minho (ULSAM), Viana do Castelo

IPD SHARING:
Plan to Share IPD: No